CLINICAL TRIAL: NCT03002350
Title: Clinical Relevance of Next-generation Sequencing Analysis for High-purity Circulating Tumor Cells From Cancer Patients With Disruptive Gene Mutation(s)
Brief Title: Clinical Relevance of NGS Analysis for High-purity CTC From Cancer Patients With Disruptive Gene Mutation(s)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Jason Chia-Hsun Hsieh, Director,Hematology&Oncology, Principal Investigator, Chang Gung Memorial Hospital
Other Study IDs: CTCNGS001; MOST-105-2314-B-182A-030 - (Other: Grantor or Funder MOST-105-2314-B-182A-030 -)
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Recurrence; Metastasis; Death
Keywords: Circulating tumor cells (CTCs); Optically induced dielectrophoresis (ODEP); Cell sorting; Next-generation sequencing (NGS); disruptive mutation
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis; Death; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — genomic DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Distant metastasis of cancer remains the major cause of cancer death. One of the evidence is that some rare cells shed from primary tumor exist in the circulation of cancer patients, which has been proven to be related to cancer relapse and distant metastasis. The number of circulating tumor cells (CTCs) or the expression status of specific marker(s) on them also correlated with the disease prognosis and treatment effects, which might change the decision of treatments. In recent years, as specific disruptive genes were discovered, such as epidermal growth factor receptor (EGFR) in non-small cell lung cancer,Kirsten rat sarcoma (KRAS) in colorectal cancer, the response rate to treatment, disease control and survival have been much improved. However, the molecular information obtained from cancer tissue depends on repeated biopsies, which is very risky and invasive to cancer patients. By means of the advances of CTCs sampling technique with genetic analysis, repeated follow-up for specific gene profiles is possible. However, the protocol has not been well-established and mature, even the correlation between primary cancer tissue and CTCs remains unknown. To tackle the problems above, the aims of the project is to isolate high-purity CTCs by the optically induced dielectrophoresis (ODEP)-based device or other cell sorting techniques and transfer to next-generation sequencing (NGS) analysis for specific disruptive genes. In the first year of the project, the investigator will testify and stabilize the platform utilizing healthy donors' blood and cancer cell lines and adjust the detailed experiment conditions. In the following year, the investigator will enroll newly diagnosed metastatic cancer patients with the disruptive gene mutation(s) and follow up the events under gene-based therapy. Comparison of NGS information between cancer tissue and CTCs will be also made as one of the major endpoints. In brief, the investigator expect the study could establish a practical method to get genetic information, to reduce the risk of re-biopsy and to achieve the ultimate goal of precision medicine.

DETAILED DESCRIPTION:
(A) Establish a High-purity isolation of CTCs to NGS platform within one year

(B) Design a Prospective trial (CTCNGS01 at www.clinicaltrials.gov) utilizing the developed technique to elucidate the baseline CTC-NGS information to cancer tissue NGS.

ELIGIBILITY:
Inclusion Criteria:

I. Age at diagnosis ≥ 20 years, II. Can fully understand the purpose of the study, pros/cons of entering the trial with clear and free mind III. With acceptable laboratory data for receiving anti-cancer therapy, adjusted by clinicians.

IV. Accept all the protocol procedures, including blood sampling and cancer tissue retrieve.

Exclusion Criteria:

I. Refuse to any of study protocol or procedure(s) at any time before or during the trial.

II. Patients without actionable gene alteration or mutation(s) in tissue at screening phase III. Patients who cannot tolerate anti-cancer therapy for at least 2 months should be withdrawn IV. Patients who cannot cooperate the imaging study for response evaluation of anti-cancer therapy V. Patients' tissue is too small to retrieve for NGS analysis. VI. Difficult blood sampling. VII. Clinician's judgement.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in three branch hospitals of Chang Gung Memorial Hospital, Taiwan including Keelung, Linkou, Taipei. Locally advanced or recurrent/metastatic head and neck cancer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | one year
  Measure response or progression events via all available imaging studies, including Chest-Xray, CT scans, or MRI, Positron Emission Tomography(PET)study. The relationship between CTCs number and time from CTCs checkpoint to disease progression will be analyzed.

SECONDARY OUTCOMES:
Overall survival | one year
  All causes of death would be documented and the relationship between CTCs number and time from CTCs checkpoint to death will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsun Hsieh, M.D, M.S, Principal Investigator — Division of Hematology-Oncology, Department of Internal Medicine, Chang Gung Memorial Hospital at Linkou
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan